CLINICAL TRIAL: NCT06520306
Title: A Study of Ropivacaine Combined With Different Concentrations of Methylene Blue Fascia Iliaca Block in Postoperative Analgesia, Cognition, and Hip Function Recovery in Patients Undergoing Hip Arthroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wang wanxia (Other)
Responsible Party: Sponsor-Investigator, Wang wanxia, Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ZY 0717
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Femoral Neck Disease
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dilute 0.25% ropivacaine + 20 mg methylene blue to 30 ml (Experimental)
  Interventions: Drug: Ropivacaine combined with methylene blue for iliac fascia block
- 0.25% ropivacaine + 40 mg methylene blue diluted to 30 ml (Experimental)
  Interventions: Drug: Ropivacaine combined with methylene blue for iliac fascia block
- 0.25% ropivacaine 30 ml (No Intervention)

INTERVENTIONS:
Drug: Ropivacaine combined with methylene blue for iliac fascia block — Ultrasound-guided fascia iliaca block using different concentrations of methylene blue combined with ropivacaine
  Arms: 0.25% ropivacaine + 40 mg methylene blue diluted to 30 ml; Dilute 0.25% ropivacaine + 20 mg methylene blue to 30 ml

SUMMARY:
Total hip arthroplasty (THA) is a commonly used treatment for hip lesions, but it is often accompanied by persistent pain after surgery, which obviously affects the quality of life of patients, so perfect postoperative analgesia is particularly important for the rapid recovery of patients. Peripheral nerve blocks are often used as postoperative analgesia for THA, and fascia iliaca compartment block (FICB) is the preferred nerve block for THA due to its good postoperative analgesic effect and fewer postoperative adverse reactions. However, the effect of nerve block with ropivacaine alone is short, and the postoperative analgesia time is limited, which seriously affects the patient's surgical recovery. Therefore, prolonging the postoperative analgesic time is an urgent problem to be solved by FICB, and some scholars recommend the combined use of local anesthetic adjuvants to prolong the block time, which is an effective and safe method. In this study, a long-acting analgesic drug, methylene blue, was selected as an adjuvant for ropivacaine for FICB, but there was no unified clinical standard for the postoperative analgesic concentration of methylene blue.

ELIGIBILITY:
Inclusion Criteria:

* Hip replacement surgery is indicated
* ASA Class II - Class III
* No history of analgesic or local anesthetic allergy
* No history of alcohol abuse or narcotic drug abuse
* Patients and their families have given informed consent and signed the informed consent form

Exclusion Criteria:

* Patient or family refusal to participate in the study
* Severe coagulation abnormalities
* Local anesthetic allergy
* Severe psychiatric illness or other communication disorder
* There is an infection at the puncture site

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale（VAS） | The first, third, and seventh days after the surgery
  Use a swimming ruler about 10 cm long, marked with 10 ticks on one side, and "0" and "10" at each end. A score of 0 indicates no pain, a score of 10 indicates the most severe pain that is unbearable, and the higher the score, the greater the degree of pain
Mini-Mental State Examination (MMSE) | Seventh day after surgery
  An examination tool to assess cognitive status
Harris Hip Scoring System | On the seventh day after surgery
  Harris (1969) proposed a scoring system to evaluate the functional status and postoperative efficacy of patients with artificial hip arthroplasty

SECONDARY OUTCOMES:
Number of postoperative salvage analgesia | From the end of the surgery to the seventh day after the surgery
Walking distance for the first time getting out of bed | From the end of the surgery to the seventh day after the surgery
Number of exercises to get out of bed within 7 days of surgery | From the end of the surgery to the seventh day after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Yang, Taizhou, China